CLINICAL TRIAL: NCT00128440
Title: A Randomized, Multiple-dose, Double-Blind, Crossover Study to Compare the Efficacy and Safety of 200 μg and 400 μg of BEA 2180 BR to Tiotropium 5 μg and Placebo When Each is Delivered by the Respimat® Inhaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: High Dose Trial in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1205.6
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: BEA 2180 BR
Drug: tiotropium

SUMMARY:
The primary objective of this study was to compare the efficacy and safety of 200 μg and 400 μg of BEA 2180 BR to tiotropium 5 μg and placebo when each was delivered by the Respimat® Inhaler once daily for four weeks in patients with COPD.

ELIGIBILITY:
1. Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 >=30% and <= 60% of predicted normal and FEV1 <=70% of FVC at the baseline PFTs at Visit 1 (at both timepoints).
2. All patients must have an increase in FEV1 of at least 12% from baseline (th e -10 minute measurement) 45 min after inhalation of 80 ?g Atrovent MDI.
3. Male or female patients 40 years of age or older.
4. Smoker or ex-smoker with a history of more than 10 pack years.

1. Patients with any other significant disease will be excluded. 2. Patients with a history of asthma or allergic rhinitis will be excluded.

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Trough forced expiratory volume (FEV1) response | baseline to 24 hours post drug administration
forced expiratory volume in one second (FEV1) area under curve 3 to 6 hours (AUC0-6h) after four weeks of treatment. | after 4 weeks

SECONDARY OUTCOMES:
Trough FVC response after 4 weeks | after 4 weeks
FEV1 and FVC peak response after 0 and 4 weeks | after 0 and 4 weeks
FVC AUC0-6h after 0 and 4 weeks | after 0 and 4 weeks
Individual FEV1 and FVC measurements at each time point | 4 weeks
Weekly mean pre-dose morning and evening PEFR | 4 weeks
Weekly mean number of occasions of rescue therapy used per day [as occasion requires (PRN) albuterol] | 4 weeks
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest | 4 weeks
Physician's Global Evaluation | 4 weeks
All adverse events | 28 weeks
Pulse rate and blood pressure (seated) recorded in conjunction with spirometry for the first three hours following dosing | 28 weeks
12-lead ECGs at baseline (-10 minutes) and at 25 minutes, 2 and 6 hours post dose on Day 1 and 29 of each treatment period (Visits 2-9) | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator
Locations (13):
- United States (13):
  - Boehringer Ingelheim Investigational Site, Lakewood, California
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - Boehringer Ingelheim Investigational Site, Pembroke Farms, Florida
  - Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - Boehringer Ingelheim Investigational Site, Reno, Nevada
  - Boehringer Ingelheim Investigational Site, Larchmont, New York
  - Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - Boehringer Ingelheim Investigational Site, Harker Heights, Texas
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - Boehringer Ingelheim Investigational Site, Tacoma, Washington